CLINICAL TRIAL: NCT01969032
Title: Phase 2 Study of Two Consequent Chemotherapy Regimens as Induction Preoperative Therapy for Patients With Locally Advanced Triple Negative Breast Cancer
Brief Title: Induction Preoperative Chemotherapy for Patients With Locally Advanced Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mona Frolova, Senior Research Associate of Department of Clinical Pharmacology and Chemotherapy, Russian Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LATN-2ICR
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Paclitaxel; Carboplatin; Doxorubicin; Cyclophosphamide; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 consequent anthracycline-taxane based chemotherapy regimens (Experimental): Paclitaxel 60 mg/m2 IV weekly plus Carboplatinum AUC2 IV weekly for 9 weeks, then Doxorubicin 25 mg/m2 IV weekly plus Endoxan 50 mg per os q.i.d. plus Capecitabine 500 mg t.i.d for 9 weeks
  Interventions: Drug: Paclitaxel, Carboplatinum, Doxorubicin, Endoxan, Capecitabine

INTERVENTIONS:
Drug: Paclitaxel, Carboplatinum, Doxorubicin, Endoxan, Capecitabine — Paclitaxel 60 mg/m2 IV weekly plus Carboplatinum AUC2 IV weekly for 9 weeks, then Doxorubicin 25 mg/m2 IV weekly plus Endoxan 50 mg per os q.i.d. plus Capecitabine 500 mg t.i.d for 9 weeks

SUMMARY:
The purpose of this study is to increase survival of patients with locally advanced triple-negative breast cancer using two consequent induction preoperative chemotherapy regimens.

DETAILED DESCRIPTION:
Compared to other breast cancer subtypes, patients with triple-negative breast cancer have a lower recurrence-free and overall survival, regardless of disease stage at diagnosis. That's why new approaches to treatment of this aggressive breast cancer subtype are extremely anticipated.

One of the ways to improve the results of treatment of locally advanced triple-negative breast cancer is intensification of induction preoperative chemotherapy regimens. Elevation of the rate of pathological complete responses after completion of intensification induction preoperative chemotherapy enables to decrease the stage and increase survival of this aggressive breast cancer subtype. We hope to achieve more clinical and pathological treatment responses than with standard chemotherapy regimens and therefore to improve treatment outcomes of this extremely adverse group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, age ≥18 years≤75
* Histologically confirmed invasive ER-, PR-, and HER2-negative (triple-negative) adenocarcinoma of the breast
* Stages Т2-4 N 2-3 M0
* Signed inform consent

Exclusion Criteria:

* Previous treatment for this breast cancer
* History of malignancy treated with curative intent within the previous 5 years with the exception of skin cancer, cervical carcinoma in situ, or follicular thyroid cancer. Patients with previous invasive cancers (including breast cancer) are eligible if the treatment was completed more than 5 years prior to initiating current study treatment, and there is no evidence of recurrent disease
* Pregnancy or breast-feeding
* Serious concurrent diseases or conditions that may alter chemotherapy conduction

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-08; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The pathological complete response rate to two consequent induction preoperative chemotherapy regimens | After 18 weeks of induction chemotherapy

SECONDARY OUTCOMES:
Disease-free survival | 3 years

OTHER OUTCOMES:
Number of patients with 3/4 Grade CTC adverse events to assess toxicity and tolerability of the chemotherapy regimens | After 18 weeks os induction chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Russian Cancer Research Center named after N.N.Blokhin RAMS, Moscow, Russia

REFERENCES:
- See also: Paclitaxel, Carboplatinum, Doxorubicin, Endoxan, Capecitabine — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: Triple Negative Locally Advanced Breast Cancer, Induction Chemotherapy — http://www.ncbi.nlm.nih.gov/pubmed